CLINICAL TRIAL: NCT03874390
Title: Effects of Ozone Therapy Adjunct to Initial Periodontal Therapy on Clinical Parameters and Inflammatory Cytokines in Chronic Periodontitis Patients
Brief Title: Effects of Ozone Therapy on Clinical Parameters and Inflammatory Cytokines in Chronic Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sema Nur Sevinc, research assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60078
Record Dates: First submitted 2016-05-01; First posted 2019-03-14 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Ozone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ozone therapy (Experimental): control group only treated with Initial Periodontal Therapy (IPT), test group treated with IPT an adjunct to gasesos ozone therapy.
  Interventions: Other: ozone
- initially periodontal therapy (Active Comparator): control group only treated with Initial Periodontal Therapy (IPT), test group treated with IPT an adjunct to gasesos ozone therapy.
  Interventions: Other: ozone

INTERVENTIONS:
Other: ozone — gaseous ozone was applied on periodontal pocket two times in one week.

SUMMARY:
The objective of this study is to evaluate of ozone therapy on both clinical and biochemical effects in periodontally patients.

DETAILED DESCRIPTION:
This study is evaluated clinical and biochemical effect of ozone therapy at 8 weeks in periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* non-smokers
* chronic periodontitis participants

Exclusion Criteria:

* smokers
* pregnancy or lactation
* individiuals with any systemic disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Clinical atachment level baseline | baseline (before treatment)
  Calculation as distance in millimeters from cement-enamel junction to the bottom of the pocket by Williams periodontal probe
Plaque index baseline | baseline (before treatment)
  As described by Silness&Löe 1964; The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  Scores 0: No plaque. scores 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  scores 2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  scores 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  score 0 considered good oral hygiene, score 3 bad oral hygiene habits. plaque index for a tooth=scores from 4 areas/4 plaque index individiual= scores from 28 tooth/28
Gingival index baseline | baseline (before treatment)
  As described by Löe&Silness 1963; The bleeding is assessed by probing gently along the wall of soft tissue of the gingival sulcus. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  score 0 - Normal, healthy gingival with sharp, non-inflamed margins. score 1 - Marginal gingivitis with minimal inflammation and edema at the free gingival. No bleeding on probing.
  score 2 - Moderate gingivitis with a wider band of inflammation and bleeding upon probing.
  score 3 - Advanced gingivitis with inflammation clinically reaching the mucogingival junction usually with ulceration.
  score 0 considered healty gingiva, score 3 assesed advanced gingival disease. gingival index for a tooth=scores from 4 areas/4 gingival index individiual= scores from 28 tooth/28
Bleeding on probing baseline | baseline (before treatment)
  As described by Ainamo&Bay 1975; The index is performed through gentle probing of the orifice of the gingival crevice. If bleeding occurs within 10 seconds a positive finding is recorded and the number of positive sites is recorded and then expressed as a percentage of the number of sites examined.
  bleeding present (+) absent (-) bleeding surface/all surface *100=% bleeding absent recording is equivalent to gingival index scores 0&1. bleeding present recording is equivalent to gingival index score 2&3.
  * 0: no bleeding on probing, healty gingiva
  * 100: all gingiva bleeding on probing; diseased gingiva.
Probing of depth baseline | baseline (before treatment)
  Measurement to the nearest millimeter from the gingival margin to the base of the clinical pocket by Williams periodontal probe
Biochemical outcomes baseline | baseline (before treatment)
  In this study, biochemical parametres including IL-1B, IL-6, IL-10, TNF-a, MMP-9 were measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) methods on Gingival Crevicular Fluid at baseline.

SECONDARY OUTCOMES:
Clinical attachment level after 8 weeks | 8 weeks after treatment
  Calculation as distance in millimeters from cement-enamel junction to the bottom of the pocket by Williams periodontal probe
Plaque index after 8 weeks | 8 weeks after treatment
  As described by Silness&Löe 1964; The measurement of the state of oral hygiene by Silness-Löe plaque index is based on recording both soft debris and mineralized deposits on the following teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  Scores 0: No plaque scores 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  scores 2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  scores 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  score 0 considered good oral hygiene, score 3 bad oral hygiene habits. plaque index for a tooth=scores from 4 areas/4 plaque index individiual= scores from 28 tooth/28
Gingival index after 8 weeks | 8 weeks after tretament
  As described by Löe&Silness 1963; The bleeding is assessed by probing gently along the wall of soft tissue of the gingival sulcus. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3.
  score 0 - Normal, healthy gingival with sharp, non-inflamed margins. score 1 - Marginal gingivitis with minimal inflammation and edema at the free gingival. No bleeding on probing.
  score 2 - Moderate gingivitis with a wider band of inflammation and bleeding upon probing.
  score 3 - Advanced gingivitis with inflammation clinically reaching the mucogingival junction usually with ulceration. score 0 considered healty gingiva, score 3 assesed advanced gingival disease.
  gingival index for a tooth=scores from 4 areas/4 gingival index individiual= scores from 28 tooth/28
Bleeding on probing after 8 weeks | 8 weeks after treatment
  As described by Ainamo&Bay 1975; the index is performed through gentle probing of the orifice of the gingival crevice. If bleeding occurs within 10 seconds a positive finding is recorded and the number of positive sites is recorded and then expressed as a percentage of the number of sites examined.
  bleeding present (+) absent (-) bleeding surface/all surface *100=% bleeding absent recording is equivalent to gingival index scores 0&1. bleeding present recording is equivalent to gingival index score 2&3.
  * 0: no bleeding on probing, healty gingiva
  * 100: all gingiva bleeding on probing; diseased gingiva.
Probing of dept after 8 weeks | 8 weeks after tretament
  Measurement to the nearest millimeter from the gingival margin to the base of the clinical pocket by Williams periodontal probe
Biochemical outcomes after 8 weeks | 8 weeks after tretment
  In this study, biochemical parametres including IL-1B, IL-6, IL-10, TNF-a, MMP-9 were measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) measured (pg/ml) by ELISA (Enzyme-Linked Immuno Sorbent Assay) methods on Gingival Crevicular Fluid at 8 weeks

IPD SHARING:
Plan to Share IPD: No